CLINICAL TRIAL: NCT01330875
Title: Lumbar Infiltration With Steroids - Effects on Pain Reduction
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: LINFRUZ01
Record Dates: First submitted 2011-04-05; First posted 2011-04-07 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-05

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: survey — no intervention. Only questionnaire after lumbar infiltration with steroids - effects on pain reduction

SUMMARY:
Questionnaire for patients who got a lumbar infiltration in our clinic. The patients will have to answer questions concerning their pain. (The lumbar infiltration itself is not part of this study)

DETAILED DESCRIPTION:
Questionnaire are given to patients who got a lumbar infiltration in our clinic of rheumatology. These patients will have to answer questions concerning their pain. (The lumbar infiltration itself is not part of this study).

ELIGIBILITY:
Inclusion criteria:

* Patients who got a lumbar infiltration in our clinic.

Exclusion criteria:

* Infiltration of thoracal or cervical spine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who got a lumbar infiltration in our clinic. The patients will have to answer questions concerning their pain (the lumbar infiltration itself is not part of this study).
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2010-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Pain reduction | week 1 and 3; month 3, 6, 12
  on visual analog scale

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Blumhardt, MD, Principal Investigator — University Hospital Zurich, Division of Rheumatology
Locations (1):
- University Hospital Zurich, Division of Rheumatology, Zurich, Switzerland